CLINICAL TRIAL: NCT06792071
Title: Feasibility and Efficacy of Radically Open Dialectical Behavior Therapy for Youth At Risk for Developing Severe and Enduring Eating Disorders
Brief Title: Evaluation of Radically Open Dialectical Behavior Therapy for Youth At Risk for Developing Severe and Enduring Eating Disorders
Acronym: RO-SEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Forskningsrådet för hälsa, arbetsliv och välfärd (FORTE) (Unknown); The Söderströmska-Königska Foundation (Unknown); Fonden för psykisk hälsa (Unknown)
Responsible Party: Principal Investigator, Martina Isaksson, PhD, Licensed psychologist, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RO-SEED
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Eating Disorders; Anorexia Nervosa; Anorexia Nervosa, Atypical; Feeding and Eating Disorders
Keywords: Anorexia Nervosa; Eating disorders; Radically open dialectical behavior therapy; Single-case experimental design study
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Single case experimental design study with multiple baselines. Thus, each individual is their own control.
Masking Description: Blinded randomization of baseline length is performed in blocks of three (4, 5, or 6 weeks) by a researcher or research assistant not otherwise involved with the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exposure to Radically Open Dialectical Behavior Therapy (RO-DBT) (Experimental)
  Interventions: Behavioral: Radically Open Dialectical Behavior Therapy (RO DBT)

INTERVENTIONS:
Behavioral: Radically Open Dialectical Behavior Therapy (RO DBT) — The intervention is a psychological treatment using Radically Open Dialectical Behavior Therapy (RO-DBT), consisting of individual therapy and skills training in group for approximately 22 weeks. Additionally, a parent group consisting of four sessions will be included as an adaptation to the adolescent group.

SUMMARY:
The goal of this experimental interventional study is to learn if the psychological treatment Radically Open Dialectical Behavior Therapy (RO-DBT), is feasible to conduct and provide positive effects for adolescents with eating disorders and emotional overcontrol. Participants will be those at risk for developing severe and enduring eating disorder symptoms, as they have not responded fully to previous treatment attempts.

Primary outcomes are feasibility and changes in eating disorder symptoms. Secondary outcomes are changes in unhelpful behaviors and experiences related to emotional overcontrol; including psychological inflexibility, suppression of emotions, and experience of loneliness.

The participants will undergo the treatment with RO-DBT, which include an approximately 22 week long treatment consisting of individual psychotherapy and parallel skills training in group.

DETAILED DESCRIPTION:
BACKGROUND

Eating disorders are psychiatric disorders characterized by loss of control over food intake. Eating disorders impair function, have serious health implications, and are associated with high mortality. The mortality in anorexia nervosa is especially striking, as it is one of the psychiatric disorders with the highest mortality rates. Approximately 20% of patients with eating disorders develop long lasting illness, referred to as Severe and Enduring Eating Disorders (SEED). However, research on this group is scarce, and knowledge about treatment options is extremely limited.

Clinical factors related to poor outcome in anorexia, including SEED, are low age at onset, premorbid obsessive-compulsive personality traits, and autistic traits. Further, dysfunctional emotion regulation (ER) has been identified as a transdiagnostic psychological risk factor for many psychiatric disorders, including eating disorders. Dysfunctional ER can be characterized by traits of excessive self-control and emotional inhibition (overcontrol). Some propose that dysfunctional ER, characterized by emotional overcontrol, is a core aspect of restrictive eating disorders such as anorexia. Further, research suggests that loneliness relates to ER, with ER strategies like excessive self-control and emotional overcontrol in youths being associated to an increased sense of social isolation and lower life satisfaction later in life, increasing the risk for enduring mental health problems.

Despite this, few studies have evaluated the feasibility and effect of transdiagnostic interventions that specifically address emotional overcontrol in clinical trials, with the specific aim to evaluate if this might have the potential to change a chronic course. Radically open dialectical behavior therapy (RO-DBT) is a treatment which has been developed to target emotional overcontrol, hypothesized to be an underlying cause of the development and maintenance of anorexia and other restrictive eating disorders. In previous studies, the research group has found more pronounced emotional overcontrol in patients with anorexia compared to bulimia, that adult patients with anorexia responded to psychological treatment with RO-DBT targeting overcontrol, and that the patients appreciated this focus in therapy. Further, one previous study has evaluated RO-DBT for adolescents with eating disorders in an uncontrolled study with positive results. However, more research is needed.

The aim of this study is to evaluate feasibility and effect of the psychological treatment RO-DBT for adolescents with primarily restrictive eating disorder symptoms that have not responded to previous treatments and who therefore are at risk for developing SEED.

Primary hypotheses

1. The RO-DBT treatment is feasible in an outpatient, adolescent, clinical setting.
2. After treatment with RO-DBT the patients will reduce their eating disorder symptoms, and, if underweight, regain weight.

Secondary hypotheses

1. Patients self-perceived health and positive feelings in social situations will increase during treatment.
2. Patients functional impairment, maladaptive overcontrol and experienced level of loneliness will decrease during treatment.
3. Patients comorbid symptoms of anxiety and depression will decrease during treatment.
4. Changes in eating disorder symptoms and maladaptive overcontrolled behaviors will be an effect of the intervention, i.e. they will be observable after introduction of the intervention.
5. The effects will remain at one-year follow-up.

PROCEDURE

Patients between 14 and 19 years old will be recruited from the Uppsala Child and adolescent psychiatry or the Adult psychiatry, either from the Eating disorder unit or the General psychiatry unit.

Anorexia is overrepresented among eating disorder patients with maladaptive overcontrol. However, as eating disorder symptoms often change in symptom expression over time, potential participants are not limited to those with a diagnosis of anorexia during the baseline assessment. Therefore, adolescent patients with eating disorder symptoms that have not responded fully to eating disorder treatment or who have relapsed after recovery will be provided with information about the treatment study, either by their ordinary caregiver or through advertisement in waiting rooms. Those interested can report this to their caregiver who contacts the research group, or patients can contact the research group themselves. Thereafter, the family is contacted via phone and booked for an information and evaluation sessions where additional verbal information is provided and the information to research persons is handed to the youths and their caregivers. If the participant is still interested and identified as overcontrolled, assessed with the The Overcontrolled Global Prototype Rating Scale developed by Lynch (2018), fulfill all inclusion but not exclusion criteria, he/she is invited to participate in the study. Informed consent is gathered from bort the participant and his/her caregivers. Participants should have gone through the diagnostic procedure at the Eating disorder unit during the last three months before enrollment in the study, if not, the same diagnostic procedure will be part of the study.

After treatment, participants will be interviewed regarding their experiences of the treatment.

STUDY DESIGN

The study is a single-case experimental design study with multiple baselines, where each individual serves as their own control. Participants will be randomized to baseline length. Baseline measures on 4-6 weeks before treatment will be assessed and contrasted to measures weekly during treatment. Follow-up will be conducted one year after treatment termination.

QUALITY ASSURANCE PLAN

Before the intervention, all therapists will be trained by authorized trainers in RO-DBT and will have provided RO-DBT to at least one individual patient. During the intervention, the team will be supervised by an expert-led consultation team. Adherence to treatment protocol will be assessed via therapist self-reports of session content which will be contrasted to the treatment outline recommended by Lynch (2018).

SAMPLE SIZE

In single-case studies, at least three replications are recommended to achieve generalizability. An analysis is conducted with three patients, followed by replication in three new patients, and so on. This means 3x3=9, which is the minimum number of participants recommended. Since dropouts are common in this patient group, 18 patients will be included.

STATISTICAL AND QUALITATIVE ANALYSES

Feasibility will be analyzed by presenting descriptive data on implementation success, treatment credibility/expectancy and adverse events. Treatment acceptability and satisfaction will be assessed by interviewing participants, and the transcripts of these interviews will be analyzed using thematic analysis..

Quantitative, repeated, data will be analyzed visually and statistically according to recommendations for single-case research. Symptoms measured weekly during a baseline before treatment (phase A) will be contrasted to weekly ratings during treatment (phase B) for each participant. For the visual analyses, the steps outlined by Kratochwill and colleagues (2013) will be followed, which include examining the level, trend, variability, immediacy of effect, overlap, and consistency of data patterns. For statistical analyses, Tau-U will be utilized as a measure of effect size. Multiple baselines between individuals will be analyzed to control for time-effects.

Within-group analyses will be calculated for the measures before treatment, after treatment, and at one-year follow-up. Reliable change index will be calculated to assess whether the changes are statistically significant and meaningful.

ELIGIBILITY:
Inclusion Criteria:

* Being 14-19 years old
* Primarily restrictive eating disorder symptoms that remain despite at least one previous treatment attempt.
* Problems related to maladaptive overcontrol
* Written informed consent (for minors, this includes consent from all caregivers and the minors themselves).

Exclusion criteria:

* Eating disorders symptoms in need of emergency care
* High risk for suicide
* An inability to respond to the questionnaires or participate in the skills class, e.g., due to lack of knowledge in Swedish.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in eating disorder symptoms measured with Eating disorder Examination Questionnaire (EDE-Q) | At baseline measurement 1 (4-6 weeks before treatment initiation), at treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely, and 6 months after the end of treatment.
  EDE-Q is a 28-item self-report questionnaire, designed to assess the range, frequency and severity of behaviors associated with an eating disorder. It is categorized into four sub-scales: Restraint, Eating Concern, Shape Concern and Weight Concern, and an overall global score. The score is obtained by calculating the mean for the total score and the subscales respectively (min = 0, max =6), higher scores indicate more severe eating disorder symptoms.
Change in eating disorder symptoms measured with Eating disorder symptom list (EDSL) | Once each week during the baseline phase (4-6 weeks before the treatment is initiated), once each week during the treatment phase (approximately 24 weeks), and at one timepoint 6 months after the end of treatment.
  The EDSL is an eight-item self-rating questionnaire designed to assess eating disorder symptoms important for diagnosis. The scale is developed to detect change, or lack of change, during treatment. Participants are asked how many days during the preceding week they: restricted the amount of food, restricted the type of food, binged, vomited, used laxatives/diuretics, exercised excessively, experienced fear of gaining weight, or had thoughts about weight and shape that affected their self-image. Responses are given on an eight-point Likert scale ranging from 0 (no days) to 7 (seven days). Higher scores indicate greater difficulties
Change in body mass index (BMI) | Once each week during the baseline phase (4-6 weeks before the treatment is initiated), once each week during the treatment phase (approximately 24 weeks), and at one timepoint 6 months after the end of treatment.
  Weight and height will be combined to report BMI in kg/m^2, assessed with a valid and reliable device in a standardized procedure. BMI is only an outcome for those with an underweight before study start, defined as 85% of expected body weight in relation to the participants age and gender.
Feasibility - treatment credibility and expectancy | At baseline measurement 1 (4-6 weeks before treatment initiation)
  The Credibility/Expectancy Questionnaire (CEQ) is a psychological assessment tool designed to measure participants' expectations of treatment effects and their perceptions of the credibility of a psychological intervention. The CEQ helps researchers understand how expectations may influence treatment outcomes. The scale consists of six items, four of them are recorded using a nine-point Likert scale, ranging from 1 (not at all) to 9 (very much), higher scores indicate a greater credibility/expectation. The scale also contains two items asking for a percentage rating of how great improvement they think/feel will happen.
Feasibility - acceptability | Within 1 month after treatment completion (on average 26 weeks after treatment initiation), or within 1 month after the participant decides to end therapy prematurely.
  Acceptability will be assessed via a qualitative interview where participants are asked to share their experiences of the treatment.
Feasibility - inclusion rates | Before first baseline, during recruitment (typically within one month before enrollment)
  Inclusion rates will be assessed by contrasting the number of participants who show interest and are evaluated for participation to the number of participant actually enrolled.
Feasibility - drop-out rates | At treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely.
  Drop-out rates will be assessed by contrasting the number of individuals who completed the treatment as planned and recommended with the number of those who dropped out prematurely, either by their own choice or due to adverse events that prevented completion.
Feasibility - Completion of homework | Once each week during the treatment phase immediately after the individual therapy session (approximately 24 weeks).
  Completion of homework will be assessed by the individual therapist rating the level of completed homework on a 3-item Likert scale: 1 (not at all completed), 2 (partially completed), and 3 (completed).
Feasibility - attendance to sessions | Once each week during the treatment phase immediately after the individual therapy session (approximately 24 weeks).
  Attendance to sessions will be calculated by contrasting the number of completed individual therapy sessions and skills sessions respectively with the expected number of completed individual therapy sessions (22-24) and skills sessions (20).

SECONDARY OUTCOMES:
Change in Eating disorder related functional impairment measured with the Clinical Impairment Assessment questionnaire (CIA) | At baseline measurement 1 (4-6 weeks before treatment initiation), at treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely, and 6 months after the end of treatment.
  The CIA is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features, Each item is rated on a four-point Likert scale ranging from 'Not at all' to 'A lot'. The minimun score is zero and the maximum score is 48, with higher scores indicating a more severe impairment.
Change in functional impairment measured with Uppsala scale of Functional Impairment in Daily life (UFID) | At baseline measurement 1 (4-6 weeks before treatment initiation), at treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely, and 6 months after the end of treatment.
  The UFID is a Five-item, five-point Likert scale that measures functional impairment in daily life on a score between 1-5. Higher scores indicate more functional impairment.
Change in self-perceived health measured with EQ-VAS | Once each week during the baseline phase (4-6 weeks before the treatment is initiated), once each week during the treatment phase (approximately 24 weeks), and at one timepoint 6 months after the end of treatment.
  The EQ-VAS is a visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Change in maladaptive overcontrol, expressive suppression, measured with Emotion regulation questionnaire (ERQ) | At baseline measurement 1 (4-6 weeks before treatment initiation), at treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely, and 6 months after the end of treatment.
  The ERQ is a self-rating instrument designed to assess individual differences in the use of emotion regulation strategies. It is composed of ten items divided into two factors: cognitive reappraisal and expressive suppression. Participants indicate their answers on a 7-point Likert-scale ranging from 1 (total disagreement) to 7 (total agreement).
Change in maladaptive overcontrol, psychological inflexibility, is measured with The Avoidance and Fusion Questionnaire for Youth (AFQ-Y) | At baseline measurement 1 (4-6 weeks before treatment initiation), at treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely, and 6 months after the end of treatment.
  The AFQ-Y is a self-rating instrument that measures psychological inflexibility. Participants rate their level of agreement on eight items on a 5-point Likert measuring one single factor. Score range is 0-24 and higher scores indicate a higher level of psychological inflexibility.
Change in social safeness and pleasure measured with the Social safeness and pleasure scale (SSPS) | At baseline measurement 1 (4-6 weeks before treatment initiation), at treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely, and 6 months after the end of treatment.
  The SSPS is an 11-item self-rating instrument that assesses the extent to which people experience their world as safe, warm, and soothing, and how connected they feel to others. Participants indicate their answers on a five-point Likert scale, ranging from 1 (almost never) to 5 (almost all the time). Scores are added together to produce a total score in the range of 11-55, with higher scores representing higher perceived social safeness and connectedness to others.
Changes in loneliness measured with the Loneliness scale | At baseline measurement 1 (4-6 weeks before treatment initiation), at treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely, and 6 months after the end of treatment.
  The Loneliness scale is an 11-item self-rating instrument includes a 6-item emotional subscale and a 5-item social subscale. Respondents are presented with a series of statements and asked to indicate the extent to which the statement applies to their situation on a four-point Likert scale. The total score can range between 0-11 with higher scores indicating greater feelings of loneliness.
Changes in loneliness measured with the UCLA Loneliness Scale | At baseline measurement 1 (4-6 weeks before treatment initiation), at treatment completion (on average 24 weeks after treatment initiation), or immediately after the participant decides to end therapy prematurely, and 6 months after the end of treatment.
  UCLA Loneliness scale is a self-rating scale designed to measure ones subjective feelings of loneliness as well as feelings of social isolation. The scale comprises three questions that measure three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation. Participants indicate their answers on a four-point Likert scale, providing a total score between 4-16, with higher scores indicating greater feelings of loneliness.
Changes in symptoms of depression and anxiety measured with the Montgomery Åsberg Depression Scale Self-assessment (MADRS-S) | Once each week during the baseline phase (4-6 weeks before the treatment is initiated), once each week during the treatment phase (approximately 24 weeks), and at one timepoint 6 months after the end of treatment.
  MADRS-S is a 9-item widely used self-rating measure of depressive severity. The intention of the scale is to give an image of the patients current state of mind. The patient grades how he/she felt during the last three days. Items are rated on a seven-point Likert scale, providing a total score between 0-54, with higher scores reflecting greater depression severity. Item 2 assess worry/anxiety and will, except being included in the calculations above, be extracted for comparing changes in anxiety.
Changes in maladaptive overcontrol during treatment, measured with weekly ratings. | Once each week during the baseline phase (4-6 weeks before the treatment is initiated), once each week during the treatment phase (approximately 24 weeks), and at one timepoint 6 months after the end of treatment.
  Four items, rated on a 7-item Likert scale, were formulated specifically for this study to assess potential change in key features and consequences of maladaptive overcontrol during treatment. Three items (regarding social connectedness, open sharing of inner feelings, and psychological flexibility) are rated so that higher scores indicate mor adaptive behaviors, one item (regarding loneliness) is rated so that higher scores indicate greater feelings of loneliness.

OTHER OUTCOMES:
The occurrence of Adverse events | Once each week during the baseline phase (4-6 weeks before the treatment is initiated), once each week during the treatment phase (approximately 24 weeks), and at one timepoint 6 months after the end of treatment.
  Adverse events, primarily defined as worsening of mental health symptoms, weight loss, increased self-harming or suicidal behaviors, or any other unwanted experiences related to the intervention, will be assessed in a checklist by the individual therapist.
Adherence to treatment protocol (ratings by therapists) assessed with the adherence form | Once each week during the treatment phase immediately after the individual therapy session (approximately 24 weeks).
  Therapist adherence to the treatment protocol will be measured by therapist ratings for each session. The adherence form will contain a checklist of the session structure where the therapist is instructed to check the boxes of which parts were included, in addition to an own evaluation of treatment adherence, rated on a scale from 1 (=low adherence), 2 (=acceptable adherence), and 3 (=good adherence) A higher score indicate better adherence. The adherence form also include a space to write down the main theme/themes of the session content.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will not be made publicly available due to confidentiality, but can be made available upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Kratochwill, T. R., Hitchcock, J., Horner, R. H., Levin, J. R., Odom, S. L., Rindskopf, D. M., & Shadish, W. R. (2013). Single-case intervention research design standards. Remedial and Special Education, 34(1), 26-38. https://doi.org/10.1177/0741932512452794
- [Background] Baudinet J, Simic M, Griffiths H, Donnelly C, Stewart C, Goddard E. Targeting maladaptive overcontrol with radically open dialectical behaviour therapy in a day programme for adolescents with restrictive eating disorders: an uncontrolled case series. J Eat Disord. 2020 Nov 13;8(1):68. doi: 10.1186/s40337-020-00338-9. PMID 33292696
- [Background] Lynch, T. R. (2018). Radically open dialectical behavior therapy: Theory and practice for treating disorders of overcontrol. New Harbinger Publications
- [Background] Isaksson M, Ghaderi A, Wolf-Arehult M, Oster C, Ramklint M. Sharing and connecting with others - patient experiences of radically open dialectical behavior therapy for anorexia nervosa and overcontrol: a qualitative study. J Eat Disord. 2021 Mar 4;9(1):29. doi: 10.1186/s40337-021-00382-z. PMID 33663612
- [Background] Isaksson M, Ghaderi A, Ramklint M, Wolf-Arehult M. Radically open dialectical behavior therapy for anorexia nervosa: A multiple baseline single-case experimental design study across 13 cases. J Behav Ther Exp Psychiatry. 2021 Jun;71:101637. doi: 10.1016/j.jbtep.2021.101637. Epub 2021 Jan 12. PMID 33524917
- [Background] Isaksson M, Ghaderi A, Wolf-Arehult M, Ramklint M. Overcontrolled, undercontrolled, and resilient personality styles among patients with eating disorders. J Eat Disord. 2021 Apr 16;9(1):47. doi: 10.1186/s40337-021-00400-0. PMID 33863394
- [Background] Oldershaw A, Lavender T, Sallis H, Stahl D, Schmidt U. Emotion generation and regulation in anorexia nervosa: a systematic review and meta-analysis of self-report data. Clin Psychol Rev. 2015 Jul;39:83-95. doi: 10.1016/j.cpr.2015.04.005. Epub 2015 May 2. PMID 26043394
- [Background] Prefit AB, Candea DM, Szentagotai-Tatar A. Emotion regulation across eating pathology: A meta-analysis. Appetite. 2019 Dec 1;143:104438. doi: 10.1016/j.appet.2019.104438. Epub 2019 Aug 31. PMID 31479694
- [Background] Wentz E, Gillberg IC, Anckarsater H, Gillberg C, Rastam M. Adolescent-onset anorexia nervosa: 18-year outcome. Br J Psychiatry. 2009 Feb;194(2):168-74. doi: 10.1192/bjp.bp.107.048686. PMID 19182181
- [Background] Keel PK, Brown TA. Update on course and outcome in eating disorders. Int J Eat Disord. 2010 Apr;43(3):195-204. doi: 10.1002/eat.20810. PMID 20186717
- [Background] Treasure J, Duarte TA, Schmidt U. Eating disorders. Lancet. 2020 Mar 14;395(10227):899-911. doi: 10.1016/S0140-6736(20)30059-3. PMID 32171414